CLINICAL TRIAL: NCT00005437
Title: Physical Activity and Cardiovascular Risk in Black Girls
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 4365; R29HL047659 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Obesity

SUMMARY:
To conduct a longitudinal study investigating the physical activity patterns, the psychosocial predictors of physical activity, and the effects of physical activity changes on blood pressure and body fatness in a cohort of African-American girls, ages 11-17.

DETAILED DESCRIPTION:
BACKGROUND:

The study contributed to an underdeveloped area of research. Physical activity is recommended as a nonpharmacological means to modify hypertension and obesity, two cardiovascular risk factors. African-American women have low levels of physical activity and high rates of obesity, hypertension, and mortality from coronary heart disease, diabetes, and hypertensive diseases. In 1992, there was an absence of longitudinal data about the physical activity habits of African-American girls even though a decline in physical activity during adolescence had been reported in other subpopulations.

DESIGN NARRATIVE:

Within the framework of puberty and maturation, the study: 1) described longitudinal patterns of physical activity; 2) assessed longitudinal changes in physical activity and concomitant changes in blood pressure and body fatness; and 3) determined psychosocial predictors of changes in physical activity. The investigators hypothesized that there would be a monotonic decrease in physical activity and that psychosocial variables would predict changes in physical activity. The study population consisted of 189 sixth grade, mostly African-American, girls in Fort Bend Independent School District, Missouri City, Texas. The girls were measured for four and a half years, ages 11 or 12 at entry of the study. Anthropometry, sexual maturation, blood pressure, physical activity habits and psychosocial predictors were measured twice a year for a total of nine examinations. Data on dietary, smoking and drinking habits were collected annually. Activity patterns, psychosocial predictors and other habits were assessed by interviews and questionnaires. Sexual maturation was assessed by menarche and the Tanner stages. Skinfold and circumference measures determined body fatness and body fat distribution.

ELIGIBILITY:
No eligibility criteria

Ages: 11 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1992-02; Study Completion 1998-01

CONTACTS AND LOCATIONS:
Overall Officials: Wedell Taylor — The University of Texas Health Science Center, Houston

REFERENCES:
- [Background] Taylor WC, Yancey AK, Leslie J, Murray NG, Cummings SS, Sharkey SA, Wert C, James J, Miles O, McCarthy WJ. Physical activity among African American and Latino middle school girls: consistent beliefs, expectations, and experiences across two sites. Women Health. 1999;30(2):67-82. doi: 10.1300/j013v30n02_05. PMID 10881759
- [Background] Taylor WC, Chan W, Cummings SS, Simons-Morton BG, Day RS, Sangi-Haghpeykar H, Pivarnik JS, Mueller WH, Detry MA, Wei II, Johnson-Masotti AP, Hsu HA. Healthy Growth: project description and baseline findings. Ethn Dis. 2002 Fall;12(4):567-77. PMID 12477144